CLINICAL TRIAL: NCT07040254
Title: The Relationship Between Paternal Support, Breastfeeding Adaptation, and Breastfeeding Self-Efficacy: Evidence From a Pregnancy School
Brief Title: Paternal Support and Its Relationship With Breastfeeding Adaptation and Self-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zehra Gürsoy (Other)
Responsible Party: Sponsor-Investigator, Zehra Gürsoy, PhN(c) Lecturer, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 52
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy; Breastfeeding Education; Breastfeeding Support; Male; Parental Support
Keywords: Parental support; breastfeeding self-efficacy; breastfeeding adaptation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnant women attending the pregnancy school with their spouses (Experimental): Participants in this group attended a six-week structured pregnancy education program together with their spouses. The program included sessions on pregnancy care, labor, breastfeeding, newborn care, and postpartum health. Data on breastfeeding adaptation and self-efficacy were collected from both mothers and fathers during the postpartum period.
  Interventions: Behavioral: Father-Inclusive Antenatal Education Program
- Pregnant Women Attending the Pregnancy School Alone (No Intervention): Participants in this group attended the six-week structured pregnancy education program without their spouses. While the fathers did not participate in the program or receive any intervention, data were collected from both mothers and fathers during the postpartum period. This group served as a control to evaluate the effects of paternal involvement in antenatal education on breastfeeding outcomes.

INTERVENTIONS:
Behavioral: Father-Inclusive Antenatal Education Program — A structured six-week antenatal education program designed for pregnant women and their spouses. The program included sessions on pregnancy care, labor, breastfeeding, newborn care, and postpartum health. Fathers in the intervention group attended the program alongside their partners and were actively engaged in discussions and learning activities related to breastfeeding support. The goal was to enhance paternal awareness and involvement to improve maternal breastfeeding adaptation and both maternal and paternal breastfeeding self-efficacy. No additional materials were provided beyond the scheduled sessions.
  Arms: Pregnant women attending the pregnancy school with their spouses

SUMMARY:
This randomized controlled trial aims to evaluate the effect of paternal support on breastfeeding adaptation and breastfeeding self-efficacy among mothers attending a structured pregnancy school program. The study is conducted at Zeynep Kamil Women and Children's Diseases Training and Research Hospital in Istanbul, Türkiye, and includes pregnant women and their partners.

Participants are assigned to an experimental group (attending the program as a couple) or a control group (mother attends alone) using random allocation. Data are collected through validated self-report scales administered during the postpartum period. The primary outcomes include changes in maternal breastfeeding adaptation and self-efficacy, and paternal breastfeeding self-efficacy. This study addresses a critical gap in perinatal care by actively involving fathers in breastfeeding support and education, aiming to improve breastfeeding outcomes and promote shared parenting roles.

DETAILED DESCRIPTION:
Detailed Description This randomized controlled experimental study investigates the effect of paternal support on breastfeeding adaptation and breastfeeding self-efficacy in mothers, using a sample drawn from participants in a pregnancy school. The study is designed in accordance with ethical principles and has received institutional review board approval.

Background and Rationale:

Breastfeeding is universally recognized as the normative standard for infant nutrition due to its numerous short- and long-term benefits for both infants and mothers. According to the World Health Organization (WHO) and UNICEF, exclusive breastfeeding is recommended for the first six months of life, followed by continued breastfeeding up to two years or beyond. Despite this, global breastfeeding rates remain suboptimal. In Türkiye, exclusive breastfeeding rates are approximately 40.7% in the first six months, and only about 30% of children continue breastfeeding until age two (TDHS, 2018).

Multiple factors influence breastfeeding duration and maternal success, one of which is the presence of social and emotional support-particularly from the infant's father. Research shows that paternal attitudes and involvement significantly influence mothers' confidence and determination to breastfeed. Fathers' support in the early postpartum period contributes positively to both maternal mental health and infant care outcomes. However, fathers are often not actively included in perinatal education or breastfeeding promotion strategies, despite evidence supporting their crucial role.

Aim:

The primary aim of this study is to determine the effect of paternal support-facilitated through participation in a structured pregnancy school program-on breastfeeding adaptation and maternal/paternal breastfeeding self-efficacy.

Study Design:

This is a prospective, randomized controlled trial with a post-test-only design. The study is conducted at Zeynep Kamil Women and Children's Diseases Training and Research Hospital between September 1, 2024, and July 1, 2025. It includes mothers and fathers who participated in a six-week structured pregnancy school. The intervention includes educational sessions on pregnancy care, nutrition, labor, pain management, breastfeeding, newborn care, and postpartum recovery.

Participants are randomly assigned to experimental and control groups using a table of random numbers based on order of enrollment in the pregnancy school. Couples who attend sessions together are assigned to the experimental group, while those where only the mother attends are assigned to the control group.

Participants:

Inclusion criteria include:

Women aged 18-49 and men aged 18-64 Residing in Istanbul and able to attend in-person sessions No mental or physical disability Ability to use smartphones or communication apps Voluntary participation with informed consent

Sample Size:

A total of 152 individuals (76 couples) are planned, with at least 38 couples per group, based on power analysis (90% power, α = 0.05).

Data Collection Tools:

Demographic Information Form: Gathers socio-demographic and pregnancy-related data.

Postpartum Breastfeeding Self-Efficacy Scale-Short Form: 14-item, 5-point Likert scale assessing mothers' confidence in breastfeeding; validated in Turkish.

Breastfeeding Adaptation Scale: 27-135 point scale with 8 subdimensions evaluating mothers' adaptation to breastfeeding; validated in Turkish.

Paternal Breastfeeding Self-Efficacy Scale-Short Form: 14-item scale assessing fathers' perceptions and support related to breastfeeding.

All instruments have received permission for use and are validated for the Turkish population.

Procedure:

First Interview: Conducted with pregnant couples upon enrollment in the pregnancy school. Those attending with their partners are assigned to the experimental group. Initial informed consent is obtained.

Second Interview: Conducted during the postpartum period, approximately four weeks after birth. Mothers and fathers complete the relevant forms.

A pilot study with 10 participants is conducted prior to full-scale data collection.

Expected Outcomes:

The study aims to demonstrate that paternal participation in perinatal education positively affects both mothers' breastfeeding adaptation and self-efficacy, and fathers' self-efficacy in supporting breastfeeding. It is anticipated that structured, father-inclusive education will improve breastfeeding outcomes and reinforce gender-equitable caregiving roles in the postpartum period.

Significance:

This study fills a significant gap in breastfeeding support strategies by actively involving fathers through a targeted educational intervention. It contributes to the broader goal of promoting sustainable breastfeeding practices and aligns with global and national public health objectives.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women aged 18 to 49 years enrolled in a pregnancy school. Male partners of the enrolled pregnant women, aged 18 to 64 years. Residing in Istanbul during the study period. Able to participate in face-to-face interviews. Able to understand and speak Turkish. Able to communicate via telephone and use digital platforms (e.g., WhatsApp, Telegram, email).

No physical or mental disability. Willing to participate and provide signed informed consent.

Exclusion Criteria:

Presence of any physical or mental disability. Unwillingness to participate in the study. Irregular attendance in pregnancy school sessions. Prior participation by either partner in the same pregnancy education program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Postpartum Breastfeeding Self-Efficacy Scale-Short Form | 4 week
  This scale was developed by Dennis in 2003 to assess breastfeeding self-efficacy during the postpartum period and was adapted into Turkish by Aluş et al. (2008) with validity and reliability established (Tokat Aluş et al., 2010). The scale consists of 14 items on a 5-point Likert scale. There are no reverse-scored items, and total scores range from a minimum of 14 to a maximum of 70. Higher scores indicate greater breastfeeding self-efficacy. The Cronbach's alpha coefficient of the original scale was reported as 0.94.
Breastfeeding Adaptation Scale | 4 week
  This scale was developed by Sun-Hee Kim (2009) to evaluate adaptation to breastfeeding. The Turkish version was validated by Dinçel and Özdilek (2021). It is a 5-point Likert-type scale consisting of 8 subdimensions. Total scores range from 27 to 135, with higher scores indicating greater adaptation to breastfeeding. The Cronbach's alpha coefficient of the scale was reported as 0.78.
Breastfeeding Self-Efficacy Scale-Short Form for Fathers | 4 week
  This scale was developed to assess fathers' perspectives and perceived effectiveness about breastfeeding. The Turkish validity and reliability study was conducted by Kucukoglu et al. (2022). The scale is self-reported, unidimensional, and consists of 14 items rated on a 5-point Likert scale. There are no reverse-scored items, and total scores range from 14 to 70. Higher scores indicate greater paternal breastfeeding self-efficacy. The Cronbach's alpha coefficient of the scale was reported as 0.93.

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Women and Children's Diseases Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to institutional policy, the data cannot be shared. The findings will be published in the related scientific article.